CLINICAL TRIAL: NCT02728609
Title: An Analysis of Cytokine Concentration in Open Abdominal Closure of Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy C. Fabian, M.D., MD, Harwell Wilson Alumni Professor, University of Tennessee
Other Study IDs: 10-00739-FB
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Trauma
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — peritoneal fluid and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blue towel: vacuum pack device: Trauma subjects undergoing temporary abdominal closure with vacuum pack technique
  Interventions: Device: Blue towel: vacuum pack device
- ABThera abdominal closure: Trauma subjects undergoing temporary abdominal closure with the commercially available ABThera vacuum device
  Interventions: Device: ABThera vacuum device

INTERVENTIONS:
Device: ABThera vacuum device — This intervention uses a commercially available vacuum device to temporarily close the abdomen following surgery.
  Other Names: Commercially available vacuum pack closure
  Groups: ABThera abdominal closure
Device: Blue towel: vacuum pack device — This intervention uses operating room towels and the application of suction to temporarily close the abdomen following surgery.
  Groups: Blue towel: vacuum pack device

SUMMARY:
The purpose of this study is to compare the pro-inflammatory and anti-inflammatory cytokines, protein content, and white blood cell (WBC) count present in the peritoneal fluid and plasma of trauma patients who undergo one of two different methods of open abdominal closure. Following analysis of the peritoneal fluid and serum samples, comparison of the results between the two groups will be completed and correlated with the overall organ function.

DETAILED DESCRIPTION:
Elevated pro and anti-inflammatory cytokines have been implicated as markers for multi-system organ failure (MOF) and death in trauma patients. Abdominal surgery can raise the levels of these cytokines and may lead to elevated plasma levels of these inflammatory cytokines possibly leading to worsening patient prognosis. Patients in whom open abdominal closure is required are often the sickest of trauma patients. Two different temporary abdominal closure techniques are generally used at the Presley Memorial Trauma Center, one using the blue towel: vacuum pack technique and one using the commercially available ABThera vacuum device from Kinetic Concepts, Inc (KCI). This study is being conducted to determine if the ABThera temporary closure technique removes a greater amount of cytokines from the abdominal cavity possibly lessening the amount of systemic or plasma cytokines and thus decreasing the incidence of MOF and death in this very ill population of patients. Additionally, this study is being conducted to determine if the white blood cell count may be lower in patients with the least cytokine values and to also investigate protein loss in these patients. The depletion of body stores of protein due to an open abdomen has great nutritional and, therefore, healing implications.

Enrollment will include 40 subjects meeting eligibility criteria into this study. The study population will include 20 patients who were temporarily closed using the ABThera device and 20 who were temporarily closed using the blue towel: vacuum pack technique. Peritoneal fluid and blood will be collected in eligible subjects immediately upon arrival to the ICU following surgery and at 12, 24, 48 and 72 hours following placement. Peritoneal fluid will be collected from the drainage system into a Lukens trap. Blood will be collected from an existing intravenous or arterial line. The peritoneal fluid will be centrifuged, separated, and frozen at -80 degrees centigrade for analysis of cytokine/inflammatory markers, protein, and WBC count. The blood specimens will be centrifuged, separated, and frozen for cytokine/inflammatory marker analysis. Chemistry and hematology values completed as standard of care will be collected from the hospital chart along with general demographics, description of injuries, treatment modalities, and outcomes.

The first samples of blood and peritoneal fluid will be obtained immediately on arrival in the ICU when other labs are being drawn as standard of care. These samples will be put aside until consent can be obtained from the legally authorized representative or the subject himself. If the research subject and/or his legally authorized representative decide that the subject should not participate in the study, the sample will be destroyed and no additional study procedures will be obtained. If the legally authorized representative is not available within 12 hours of the initial specimen and the subject is unable to consider participation within 12 hours of the initial specimens, the subject will not be enrolled into the study, and samples obtained immediately on arrival to the ICU will be destroyed.

After all analyses are completed, comparison of the cytokine levels, WBC count, and protein extraction between the two vacuum methods will be completed and correlated to the patients' overall organ function.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age who have been admitted following abdominal trauma and require open laparotomy
* Those who are closed using either the blue towel: vacuum pack method or the ABThera vacuum device
* Those who can be enrolled within 12 hours of placement of temporary abdominal closure

Exclusion Criteria:

* Those who cannot give informed consent and do not have a Legally Authorized Representative available
* Prisoners are excluded
* Pregnant women are excluded
* Those under 18 years of age and older than 75 years of age
* Those who do not require temporary abdominal closure using either the blue towel: vacuum pack technique or with the ABThera vacuum device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Presley Memorial Trauma Center undergoing open abdominal closure with a vacuum device will be invited to participate. A total of 40 patients with 20 patients in each group will be included.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in cytokine levels over 72 hours in peritoneal fluid in each enrolled subject | Change in cytokine levels over 72 hours following placement of the device
  Fluid will be obtained from the collection portion of the device into a Lukens trap. Fluid will be centrifuged into separate specimens and frozen at -80 degrees centigrade prior to analysis. Specimens will be analyzed using standard laboratory process.

SECONDARY OUTCOMES:
Change in white blood cell count in peritoneal fluid over 72 hours following placement of the device in each enrolled subject | Serial samples obtained over 72 hours following placement of the device
  Fluid will be obtained from the collection portion of the device into a Lukens trap. Fluid will be centrifuged into separate specimens and frozen at -80 degrees centigrade prior to analysis. Specimens will be analyzed using standard laboratory process.
Change in protein content in peritoneal fluid over 72 hours following placement of the device in each enrolled subject | Serial samples obtained over 72 hours following placement of the device
  Fluid will be obtained from the collection portion of the device into a Lukens trap. Fluid will be centrifuged into separate specimens and frozen at -80 degrees centigrade prior to analysis. Specimens will be analyzed using standard laboratory process.
Change in cytokine levels in serum samples over 72 hours following placement of the device in each enrolled subject | Serial samples obtained over 72 hours following placement of the device
  Serum samples will be collected for an indwelling intravenous catheter, centrifuged into separate specimens and frozen for cytokine/inflammatory marker analysis. Specimens will be analyzed using standard laboratory process.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C. Fabian, MD, Principal Investigator — University of Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spindler-Vesel A, Wraber B, Vovk I, Kompan L. Intestinal permeability and cytokine inflammatory response in multiply injured patients. J Interferon Cytokine Res. 2006 Oct;26(10):771-6. doi: 10.1089/jir.2006.26.771. PMID 17032171
- [Background] Kowal-Vern A, Ortegel J, Bourdon P, Chakrin A, Latenser BA, Kimball D, Casey LC. Elevated cytokine levels in peritoneal fluid from burned patients with intra-abdominal hypertension and abdominal compartment syndrome. Burns. 2006 Aug;32(5):563-9. doi: 10.1016/j.burns.2005.12.010. PMID 16766124
- [Background] Liener UC, Bruckner UB, Knoferl MW, Steinbach G, Kinzl L, Gebhard F. Chemokine activation within 24 hours after blunt accident trauma. Shock. 2002 Mar;17(3):169-72. doi: 10.1097/00024382-200203000-00002. PMID 11900333